CLINICAL TRIAL: NCT01026948
Title: Feasibility and Acceptability of the Combination of Propess and AN24 Monica for Outpatient Labour Induction (PRAM)
Acronym: PRAM
Status: Completed | Type: Observational
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: LWH0764
Record Dates: First submitted 2009-12-03; First posted 2009-12-07 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2011-11

CONDITIONS: Intrapartum Fetal Monitoring; Pregnancy
Keywords: Induction of labour; Intraprtum fetal monitoring
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Propess and Monica AN24 care package: Women who are eligible and consent to recruitment will receive the Propess and Monica AN24 care package for outpatient induction of labour
  Interventions: Drug: Dinoprostone; Device: Monica AN 24

INTERVENTIONS:
Drug: Dinoprostone — Propess© vaginal delivery system consists of a non-biodegradable polymeric drug delivery device containing 10 mg Dinoprostone (PGE2) dispersed throughout its hydrogel matrix. The retrieval vaginal insert expands to twice its size and releases a continuous and predictable dose of Dinoprostone at a rate of approximately 0.3 mg/hr over 24 hours (4-5 mg PGE2 over 12 hours) in women with intact membranes whereas release is higher and more variable in women with premature rupture of membranes.
  Other Names: Propess
Device: Monica AN 24 — AN24 Monica is a portable, battery powered device designed to passively monitor a pregnant mother and unborn baby. The device is attached via a suitable cable assembly which in turn attaches to 5 standard disposable electrodes placed on the abdomen of a pregnant woman and is intended for use in either the home or hospital environment.
  Other Names: CE0843

SUMMARY:
In order to confirm the feasibility of home monitoring with Monica AN 24, a licensed portable device for measuring fetal and maternal electrocardiogram (ECG), and the feasibility of inpatient monitoring with Monica AN 24 in patients with Propess (a vaginal licensed drug delivery system used for induction of labour), we will perform a pilot study that will include 20 women in each arm.

Feasibility of monitoring with Monica AN 24 both in hospital and at home will be confirmed in a pilot study. The success will be defined as at least 10 minutes of continuous satisfactory trace in any given hour in at least 80% of the patient.

A main study will then be conducted to assess the feasibility and acceptability of the Propess and Monica AN24package of care for women undergoing induction of labour.

The research questions are:

1. Is outpatient induction with continuous monitoring technically feasible?
2. Does the Propess and Monica AN24 care package of care provide adequate clinical information in line with the UK National Institute of Clinical Evidence (NICE) Guideline for Induction of labour?
3. Is outpatient induction a concept that appeals to women?
4. What do women consider to be the advantages and disadvantages of this package of care?
5. What would women consider to be positive and/or negative outcome in future clinical trials of outpatient induction?
6. Do fetuses with abnormal electrocardiogram (ECG) patterns have evidence of subclinically impaired cardiac function (feasibility study)?
7. Do elevated concentrations of white blood cell components in the umbilical cord blood at birth influence fetal electrocardiogram (feasibility study)?

DETAILED DESCRIPTION:
Inclusion criteria

Women with singleton pregnancy and cephalic presentation booked for induction of labour with unfavourable cervix (Bishop score <6) and normal pre-induction fetal monitoring.

Low risk women in the context of this study include:

* Uncomplicated pregnancy requiring induction of labour after completed 37 weeks of of pregnancy with normal fetal assessment including:

  1. Social inductions/maternal requests
  2. Induction of labour for symphysis pubic dysfunction
  3. Obstetric Cholestasis
  4. Nonspecific Proteinuria (without any other medical problems)
* Parity < 4
* Intact membranes at study entry
* Living within a reasonable distance from the hospital (i.e., not more than approximately 60 minutes driving time)
* Caregiver present at all times while at home
* Easy access to a safe method of transport for return to hospital
* Easy access to a telephone (either land line or mobile with good service)
* Agrees to remove the pessary herself following instructions in the patient leaflet
* Written informed consent

Exclusion criteria

* Previous caesarean section
* Abnormal preinduction Cradiotocogram (CTG)
* Multiple pregnancy
* Fetal malformation or chromosomal abnormality
* Maternal age less than 18 years
* Contraindication to Propess induction
* Breech Presentation
* Foetal growth restriction
* Hypertension
* All Diabetics

Recruitment

In Liverpool Women's Hospital, women who have completed 37 weeks of Pregnancy and require induction of labour (as per inclusion/exclusion criteria above) while attending Antenatal clinic, delivery suite or the Obstetric Assessment Unit are offered management options. Women who have normal cardiotocogram (CTG), normal amniotic fluid volume and cephalic presentation confirmed by ultrasound, and who decide to have induction of labour will be approached by one of the investigators. The participant information sheet will be given to the woman, and participation in the study offered.

Women who accept participation will be approached again when admitted to the Induction Suite 1-3 days later. Women who labour spontaneously before induction day will be managed according to the standard hospital protocol and will not be asked to take part in the study.

On admission to the Induction Suite the woman will be asked to sign the informed consent form and the eligibility of consenting women will be confirmed.

Study progress

Women who sign a consent form will have a Monica AN24 fetal monitor attached to the abdomen. Women will then follow the standard clinical protocol which includes:

* 30 minutes of fetal heart rate monitoring (FHR). This must be reassuring to continue with the study;
* Prescription and administration of Propess
* A further 1 hour of FHR monitoring with the woman in a recumbent position in hospital

If remote FHR monitoring cannot be established during initial assessment in the hospital, women will remain in hospital. If the in-hospital FHR signal is satisfactory, fetal monitoring will continue to be performed with Monica AN24 throughout her labour induction. If at any point the signal is deemed inadequate, standard CTG monitoring will be commenced.

Women will be invited to complete a semi-structured diary throughout the outpatient episode of care. The woman's main supporter during labour (partner, mother, or friend) will also be invited to add comments in the diary. The diary will be collected on admission to hospital and placed in an opaque envelope. The diary will be collected by the Qualitative Team and will not be read by the clinicians/researchers involved in the clinical care.

Women who meet all of the inclusion and none of the exclusion criteria and with a satisfactory in-hospital Monica AN24 signal will be taken through the instruction leaflets for the AN24 and Propess. If they are comfortable with both sets of instructions and the staff member believes they understand the study and how to handle an emergency situation, they will be allowed home. They will be advised that in case of research staff observing a suboptimal/non-reassuring fetal heart rate signal, they will be contacted by phone to come back to the hospital. Participating women will also be provided with a specially enabled mobile phone for the duration of their involvement with the study.

The patient leaflets provided to women who are deemed suitable for home monitoring will include instructions to contact hospital staff and come back to the hospital in case of:

1. vaginal bleeding
2. painful uterine contractions requiring pain relief
3. rhythmic, firm, uterine contractions occurring at a frequency of ≥ 3 in 10 minutes and lasting 45 seconds or more
4. rupture of membranes
5. Pessary falling out

Women will be provided with the contact number for the Induction Suite (staffed 24/7), and they may contact the Induction Suite staff by telephone for reassurance at any time.

The Monica AN24 monitoring will upload data to the central data base every 30 seconds via Bluetooth technology. The fetal heart rate and uterine activity pattern will be displayed on the PC monitor situated on the Induction Suite. This will be reviewed periodically by an experienced midwife as per standard hospital practice for women undergoing cervical ripening.

Women will be told to return to the hospital in case of:

1. Evidence of uterine hypertonus defined as a single contraction with duration of at least 2 minutes
2. Evidence of uterine tachysystole defined as at least 6 contractions in 10 minutes for 2 consecutive 10 minute periods
3. Non reassuring/pathological fetal heart rate (FHR)
4. In case of regular uterine contractions (at least 3 in 10 minutes) the patient will be contacted by the midwife and asked if the contractions are painful. If the patient refers the contractions as non painful, home monitoring will be continued.

Whilst the participant is at home, should a situation arise that the staff believes requires removal of the pessary (Propess), they will telephone the participant and instruct her to remove and dispose of the insert, and request that she should immediately return to the hospital. The staff member evaluating the situation will also determine whether emergency transport is required, i.e., ambulance, or whether car/taxi is acceptable.

At 24 hours, assuming none of the above reasons for returning to hospital has occurred; women will be asked to return to hospital for removal of pessary and further assessment. Further management will be according to the standard hospital protocol for failed induction.

Provided that the FHR signal from the Monica AN24 device is adequate, the device will be used for monitoring throughout the first stage of labour. In the second stage of labour a standard cardiotocogram (CTG) monitoring will be added.

If at any point of the labour the signal is considered inadequate, standard cardiotocogram (CTG) monitoring will be provided.

After birth, cord blood will be collected for analysis of lactates, cardiac enzymes, interleukin-6 (IL-6) and reactive protein C. These results will not be disclosed to the clinicians and will not influence subsequent management. Women will also be asked to give consent (optional) for one neonatal electrocardiogram (ECG) recording before hospital discharge if feasible.

Women will also be asked to participate in a face to face interview after birth to determine their views on the outpatient care. This interview will be arranged by a member of the Qualitative Team after discharge from hospital and take place either at home or at hospital depending on the woman's wishes.

ELIGIBILITY:
Inclusion criteria

Women with singleton pregnancy and cephalic presentation booked for induction of labour with unfavourable cervix (Bishop score <6) and normal pre-induction fetal monitoring.

Low risk women in the context of this study include:

* Uncomplicated pregnancy requiring induction of labour after completed 37 weeks of of pregnancy with normal fetal assessment including:

  1. Social inductions/maternal requests
  2. Induction of labour for symphysis pubic dysfunction
  3. Obstetric Cholestasis
  4. Nonspecific Proteinuria (without any other medical problems)
* Parity < 4
* Intact membranes at study entry
* Living within a reasonable distance from the hospital (i.e., not more than approximately 60 minutes driving time)
* Caregiver present at all times while at home
* Easy access to a safe method of transport for return to hospital
* Easy access to a telephone (either land line or mobile with good service)
* Agrees to remove the pessary herself following instructions in the patient leaflet
* Written informed consent

Exclusion criteria

* Previous caesarean section
* Abnormal preinduction cardiotocogram (CTG)
* Multiple pregnancy
* Fetal malformation or chromosomal abnormality
* Maternal age less than 18 years
* Contraindication to Propess induction
* Breech Presentation
* Foetal growth restriction
* Hypertension
* All Diabetics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In Liverpool Women's Hospital, women who have completed 37 weeks of Pregnancy and require induction of labour (as per inclusion/exclusion criteria above) while attending Antenatal clinic, delivery suite or the Obstetric Assessment Unit are offered management options. Women who have normal cardiotocogram(CTG), normal amniotic fluid volume and cephalic presentation confirmed by ultrasound, and who decide to have induction of labour were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zarko Alfirevic, Professor, Principal Investigator — Liverpool Women's NHS Foundation Trust
Locations (1):
- Liverpool Women's NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Propess and Monica AN24 Care Package: Women who are eligible and consent to recruitment will receive the Propess and Monica AN24 care package for outpatient induction of labour.
  Propess© consists of a drug delivery device containing 10 mg Dinoprostone dispersed throughout its hydrogel matrix. The retrieval vaginal insert expands to twice its size and releases a continuous and predictable dose of Dinoprostone at a rate of approximately 0.3 mg/hr over 24 hours (4-5 mg PGE2 over 12 hours.
  AN24 Monica is a portable, battery powered device designed to passively monitor a pregnant mother and unborn baby. The device is attached via a suitable cable assembly which in turn attaches to 5 standard disposable electrodes placed on the abdomen of a pregnant woman and is intended for use in either the home or hospital environment.
Period: Overall Study
Arm/Group | Propess and Monica AN24 Care Package
Started | 70
Completed | 62 (8 Women were recalled because of signal loss)
Not Completed | 8
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Arm/Group | Propess and Monica AN24 Care Package
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 70

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Defined as the Number of Eligible Women Who Are Successfully Monitored Remotely With Trans-abdominal Fetal Electrocardiogram (ECG) Monitoring Device (Monica AN24) While Undergoing Labour Induction.
Description: Outpatient induction is when women recieve medication to induce labour at the hospital, but can then go home for monitoring until labour progresses. When 'standard' Doppler Ultrasound FHR technology is used, women may feel restrained as the Doppler-FHR machine (which is bench-top device) is connected to the transducer which is then mounted on the woman's abdomen and attached by an elastic belt, which is known to be uncomfortable for pregnant woman. The AN 24 device is portable and attaches to the patients abdomen allowing remote fetal monitoring whilst the women are at home.
Time Frame: 6 months
Population: 70 women were recruited to the study, but 8 women were called back to the unit because of signal loss.
Measure: Number; unit: participants
Arm/Group | Propess and Monica AN24 Care Package
Number analyzed (Participants) | 62
participants | 62

2. Secondary Outcome: Number of Participants Who Were Satisfied With Monitoring at Home
Description: Maternal views were assessed by semi-structured diaries,recording women's ratings on a 4 point scale (very satisfied, satisfied, slightly disatisfied, very disatisfied)of how well they were coping and their satisfaction with outpatient experience.Women completed diaries at least once every two hours at home.Mean scores were calculated for women's ratings of coping, comfort satisfaction and location preference. An interpretive approach was utilised for all open responses. Comments made in the free-text spaces of diaries were categorised to contextualise women's ratings of their experience
Time Frame: 6 months
Population: 51 women out 70 returned the semistructured diaries. All the diaries were assessed as explained above.
Measure: Number; unit: participants
Groups:
- Acceptability: Maternal views were assessed using semi-structured diaries
Arm/Group | Acceptability
Number analyzed (Participants) | 51
participants | 46

ADVERSE EVENTS:
Arm/Group | Propess and Monica AN24 Care Package
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes